CLINICAL TRIAL: NCT05659069
Title: The Effect of Inferior Alveolar Nerve Lateralization on Nutritional Status, Masticatory Performance and Speech; Observational Study
Brief Title: Influence of Mandibular Nerve Lateralization on Nutrition and Speech
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MU_DHF_SBF_05
Record Dates: First submitted 2022-12-11; First posted 2022-12-21 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Alveolar Bone Loss; Bone Deformity
Keywords: Dental implants; Mandibular nerve; Nutritional status
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 10 patients with dental implant placement without inferior alveolar nerve lateralization
- Lateralization group: 10 patients with dental implant placement with inferior alveolar nerve lateralization.

SUMMARY:
This study aimed to evaluate the effects of lip numbness on the nutritional status and speech of patients who underwent inferior nerve lateralization for dental implant placement in the mandibular posterior region. For this purpose, observational follow-up of two groups of patients will be performed. The control group will include patients with standard implant placement in the mandibular posterior region. The test group will consist of patients with implant placement in the mandibular posterior region with inferior alveolar nerve lateralization. The patients will be evaluated before implant surgery and followed up for four months until the final prosthesis is placed. Changes in nutritional status, masticatory performance and speech abilities will be assessed during this process.

ELIGIBILITY:
Inclusion Criteria:

* A standard dental implant with or without lateralization of the inferior alveolar nerve in the posterior region of the mandible at the Marmara University Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery clinic.
* The patient accepted to participate in the study and gave written/verbal consent

Exclusion Criteria:

* Dental implant placement in the posterior region of the mandible with additional surgical methods (onlay/inlay graft, directed tissue regeneration, etc.) other than nerve lateralization.
* Patients had a neurosensory disorder in the maxillofacial region before implant surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with missing teeth in the posterior mandibular region and planned dental implant construction will constitute the study population.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in a neurosensory disturbance with a two-point discrimination test | Baseline function evaluation, followed by reevaluations at 7th days, 2, 3 months.
  Using a calliper, this test will be carried out. Care should be given to ensure that both calliper tips are touching the lower lip simultaneously until the patient can distinguish between two points of contact, at which point the distance between the two points is noted.
Change from baseline in lip sensitivity pattern with semmes-weinstein monofilament test | Baseline function evaluation, followed by reevaluations at 7th days, 2, 3 months.
  Mapping of the Semmes-Weinstein monofilament pressure thresholds in the lower lip's predetermined regions.
Change from baseline in nutritional status | Baseline evaluation, followed by reevaluations at 7th days, 2, 3 months.
  The Subjective Global Assessment (SGA) will be used to assess changes in nutritional status. SGA is an easy-to-apply, a low-cost and reliable method frequently used to evaluate malnutrition status. After the patient is assessed according to specific criteria, the level of malnutrition is determined by the evaluator's subjective point of view. It is a four-part evaluation. These are weight loss and food intake history, gastrointestinal system symptoms, functional capacity, metabolic requirements, and physical examination. The analysis of the information and the results from it are scored as A, B, C. If the patient is well-nourished, he is classified as A, moderately malnourished, B, and severely malnourished, C. SGA will be applied by the researchers in face-to-face meetings.
Change in acoustic characteristics of speech | Baseline evaluation, followed by reevaluations at 7th days, 2, 3 months.
  PRAAT software will be used for scientific analysis of speech and phonetics. In our study, the acoustic properties of speech will be recorded and compared with the help of PRAAT before and after the implant, and it will be examined whether these properties have changed or not. Pitch characteristics, jitter values, shimmer values, intensities and speech breaks, if any, will be observed.
  Shimmer (dB): Shimmer is a parameter that shows the relative change between the sound wave amplitudes at short intervals. The peak amplitude of each period is compared with the peak amplitude of the next period, and shimmer can be calculated in dB.
  Jitter: Jitter is the parameter that shows the variability of the vibratory cycle frequency with respect to the subsequent cycle frequency.

SECONDARY OUTCOMES:
Change from baseline in the masticatory performance | Baseline function evaluation, followed by reevaluations at 7th days, 2, 3 months.
  The masticatory performance of patients at the baseline, one month and six months later will be taken with a colour-changeable gum called "XYLITOL" (70x20x1 mm 3 g; Masticatory Performance Evaluating Gum XYLITOL, Lotte, Tokyo, Japan). Colour-changeable gum was first developed to evaluate a person's masticatory performance, changing colour as it is chewed. The gum will be chewed 60 times by the TMD patients. These values will be recorded and compared with the baseline, 1, 2, 3, and 4 months. After chewing, the gum colour will be evaluated according to the improved colour scale. The Colour scale ranges from 1-10, and the masticatory performance will be assessed as poor (1-6), average (7-8), or reasonable (9-10) with the improved colour scale.
Change from baseline in body weight | Baseline evaluation, followed by reevaluations at 7th days, 2, 3 months.
  Body weight will be evaluated during face-to-face interviews with patients in baseline, 1, 2, 3, and 4 months with the Tanita DC-360 body analyser. Patients will be asked to remove all metal items (rings, earrings, bracelets, watches, phones, etc.) and any heavy clothing, shoes, or socks before stepping on the device. The device was set to -1.0 kg for the remaining clothes.
Change from baseline in food consumption | Baseline evaluation, followed by reevaluations at 7th days, 2, 3 months.
  To evaluate the food consumption of the patients included in the study, at the baseline, 1, 2, 3, and 4 months will be taken with the 24-hour recall method. The amount of nutrients included in the meals will be calculated by using the "Standard Recipes" book, and the measurement amounts will be calculated by using the "Food Photo Catalogue" book. The data obtained from the 24-hour recall method will be analyzed using the "Computer Assisted Nutrition Program, Nutrition Information Systems Package Program (BEBIS)", and the amount of energy, carbohydrates, protein, fat, fiber and micronutrients consumed by participants will be calculated. Intake of energy, macronutrients, fiber and micronutrients will be compared with baseline evaluation followed by reevaluations.
Change from baseline in depression test | Baseline evaluation, followed by reevaluations at 7th days, 2, 3 months.
  Beck Depression Scale will be used for the evaluation of depression status. The scale consists of 21 items. Two items are divided into emotions, eleven into cognitions, two into behaviours, five into physical symptoms, and one into interpersonal symptoms. Patients will be asked to choose the most appropriate question for their situation. Each question will be scored as 0, 1, 2, or 3, and scores ranging from 0-63 will be obtained. The results will be evaluated as 0-9 none/minimal depression, 10-18 mild depression, 19-29 moderate depression, and 30-63 severe depression.
Change from baseline in observational assessment of chewing | Baseline function evaluation, followed by reevaluations at 7th days, 2, 3 months.
  Fried pieces of meat, fried chicken, peeled apples, raw carrots, almonds, hazelnuts, slices of chocolate, bread, pasta, rice, feta cheese, meatballs, boiled carrots, and boiled vegetables prepared with the same standard procedures for each patient will be presented to the patients, and their chewing will be video recorded. It will be taken. Three different researchers evaluated the video recordings; They will be categorised as (I) hard to chew, (II) slightly hard to chew, and (III) easy to chew.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krekmanov L, Kahn M, Rangert B, Lindstrom H. Tilting of posterior mandibular and maxillary implants for improved prosthesis support. Int J Oral Maxillofac Implants. 2000 May-Jun;15(3):405-14. PMID 10874806
- [Background] de Vicente JC, Pena I, Brana P, Hernandez-Vallejo G. The use of piezoelectric surgery to lateralize the inferior alveolar nerve with simultaneous implant placement and immediate buccal cortical bone repositioning: a prospective clinical study. Int J Oral Maxillofac Surg. 2016 Jul;45(7):851-7. doi: 10.1016/j.ijom.2016.01.017. Epub 2016 Feb 17. PMID 26897328
- [Background] Abayev B, Juodzbalys G. Inferior alveolar nerve lateralization and transposition for dental implant placement. Part I: a systematic review of surgical techniques. J Oral Maxillofac Res. 2015 Mar 30;6(1):e2. doi: 10.5037/jomr.2014.6102. eCollection 2015 Jan-Mar. PMID 25937873
- [Background] Alling CC. Lateral repositioning of inferior alveolar neurovascular bundle. J Oral Surg. 1977 May;35(5):419. No abstract available. PMID 265383
- [Background] Deryabin G, Grybauskas S. Dental implant placement with inferior alveolar nerve repositioning in severely resorbed mandibles: a retrospective multicenter study of implant success and survival rates, and lower lip sensory disturbances. Int J Implant Dent. 2021 Jun 9;7(1):44. doi: 10.1186/s40729-021-00334-x. PMID 34105021
- [Background] Khojasteh A, Hassani A, Motamedian SR, Saadat S, Alikhasi M. Cortical Bone Augmentation Versus Nerve Lateralization for Treatment of Atrophic Posterior Mandible: A Retrospective Study and Review of Literature. Clin Implant Dent Relat Res. 2016 Apr;18(2):342-59. doi: 10.1111/cid.12317. Epub 2015 Jun 17. PMID 26082191
- [Background] Vetromilla BM, Moura LB, Sonego CL, Torriani MA, Chagas OL Jr. Complications associated with inferior alveolar nerve repositioning for dental implant placement: a systematic review. Int J Oral Maxillofac Surg. 2014 Nov;43(11):1360-6. doi: 10.1016/j.ijom.2014.07.010. Epub 2014 Aug 12. PMID 25128261
- [Background] Palacio Garcia-Ochoa A, Perez-Gonzalez F, Negrillo Moreno A, Sanchez-Labrador L, Cortes-Breton Brinkmann J, Martinez-Gonzalez JM, Lopez-Quiles Martinez J. Complications associated with inferior alveolar nerve reposition technique for simultaneous implant-based rehabilitation of atrophic mandibles. A systematic literature review. J Stomatol Oral Maxillofac Surg. 2020 Sep;121(4):390-396. doi: 10.1016/j.jormas.2019.12.010. Epub 2020 Jan 2. PMID 31904530
- [Background] Kan JY, Lozada JL, Goodacre CJ, Davis WH, Hanisch O. Endosseous implant placement in conjunction with inferior alveolar nerve transposition: an evaluation of neurosensory disturbance. Int J Oral Maxillofac Implants. 1997 Jul-Aug;12(4):463-71. PMID 9274075
- [Background] Hirsch JM, Branemark PI. Fixture stability and nerve function after transposition and lateralization of the inferior alveolar nerve and fixture installation. Br J Oral Maxillofac Surg. 1995 Oct;33(5):276-81. doi: 10.1016/0266-4356(95)90037-3. PMID 8555142
- [Background] Lin CS, Wu SY, Huang HY, Lai YL. Systematic Review and Meta-Analysis on Incidence of Altered Sensation of Mandibular Implant Surgery. PLoS One. 2016 Apr 21;11(4):e0154082. doi: 10.1371/journal.pone.0154082. eCollection 2016. PMID 27100832
- [Background] Abayev B, Juodzbalys G. Inferior Alveolar Nerve Lateralization and Transposition for Dental Implant Placement. Part II: a Systematic Review of Neurosensory Complications. J Oral Maxillofac Res. 2015 Mar 30;6(1):e3. doi: 10.5037/jomr.2014.6103. eCollection 2015 Jan-Mar. PMID 25937874
- [Background] Tomazi MA, da Silveira Gerzson A, Neto AM, da Costa ALP. In-Block Lateralization as a New Technique for Mobilization of the Inferior Alveolar Nerve: A Technique Case Series. J Oral Implantol. 2021 Aug 1;47(4):333-341. doi: 10.1563/aaid-joi-D-20-00041. PMID 32838423
- [Background] Fernandez Diaz JO, Naval Gias L. Rehabilitation of edentulous posterior atrophic mandible: inferior alveolar nerve lateralization by piezotome and immediate implant placement. Int J Oral Maxillofac Surg. 2013 Apr;42(4):521-6. doi: 10.1016/j.ijom.2012.10.015. Epub 2012 Nov 12. PMID 23153786
- [Background] Hassani A, Saadat S, Moshiri R, Shahmirzad S, Hassani A. Nerve Retraction During Inferior Alveolar Nerve Repositioning Procedure: A New Simple Method and Review of the Literature. J Oral Implantol. 2015 Jul;41 Spec No:391-4. doi: 10.1563/AAID-JOI-D-13-00108. Epub 2013 Dec 17. PMID 24344674
- [Background] Renton T, Dawood A, Shah A, Searson L, Yilmaz Z. Post-implant neuropathy of the trigeminal nerve. A case series. Br Dent J. 2012 Jun 8;212(11):E17. doi: 10.1038/sj.bdj.2012.497. PMID 22677874
- [Background] Renton T, Yilmaz Z. Profiling of patients presenting with posttraumatic neuropathy of the trigeminal nerve. J Orofac Pain. 2011 Fall;25(4):333-44. PMID 22247929